CLINICAL TRIAL: NCT03066193
Title: Examining the Efficacy of a Therapeutic Combination of Dronabinol (Synthetic Δ9-tetrahydracannabinol) and Palmitoylethanolamide for Tourette Syndrome
Brief Title: Efficacy of a Therapeutic Combination of Dronabinol and PEA for Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Neurothera Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1610018525
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Results first posted 2019-12-19 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Tourette Syndrome
Keywords: Motor tics; Vocal tics; Cannabinoids; Dronabinol; PEA; Palmitoylethanolamide; Tourettes; TS
MeSH Terms: conditions — Tourette Syndrome; Tics | interventions — Dronabinol; palmidrol

STUDY DESIGN:
Intervention Model Description: Participants will receive two active medications and will be followed-up bi-weekly for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dronabinol and Palmitoylethanolamide (Experimental): All participants will be titrated up on Dronabinol dose during the first week of the trial (2.5mg Dronabinol for 3 days and then 5mg Dronabinol for 4 days increasing to 10mg Dronabinol for the remainder of the trial). Dronabinol will only be increased to 10mg at the week 1 assessment if the subject is tolerating the 5mg dose of Dronabinol and the Dronabinol may be reduced based on patient side-effects. All participants will receive two 400mg tablets of PEA daily for the same 12 weeks that they receive the Dronabinol.
  Interventions: Drug: Dronabinol and Palmitoylethanolamide

INTERVENTIONS:
Drug: Dronabinol and Palmitoylethanolamide — Participants will receive Dronabinol which will be slowly titrated in the first week of the study. They will be followed for a total of 12 weeks; in addition, participants will receive the PEA in a standing dose of 400mg. They will be followed for a total of 12 weeks.
  Other Names: synthetic Δ9THC; Marinol; C21H30O2; Δ9-Tetrahydracannabinol; PEA; C18H37NO2; PeaPure; N-palmitoylethanolamine; MimyX; Impulsin; Normast

SUMMARY:
This is an investigator-initiated proof of concept study with the purpose to examine the safety, tolerability and feasibility of Dronabinol (synthetic Δ9-THC) and PEA for the treatment of adults with Tourette syndrome.

DETAILED DESCRIPTION:
The investigators propose a 12-week, investigator-initiated, open-label trial of a therapeutic combination of Dronabinol and PEA in 18 adults with Tourette syndrome. Participants will receive Dronabinol and PEA in combination for the duration of the trial. The goal for this pilot study is to (1) provide initial safety, feasibility and tolerability data on both Dronabinol and PEA in a TS population and (2) provide data in order to make a more informed decision regarding the appropriate sample size and design of a larger clinical trial to prove efficacy (i.e. sample size and trial duration in large efficacy trial of the Dronabinol/PEA combination in TS).

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18-60 years of age
* Meet DSM-5 criteria for the diagnosis of Tourette syndrome
* Significant current tic symptoms: YGTSS total tic score greater than or equal to 22 at baseline
* On stable psychiatric medication regimen for a minimum of 4 weeks prior to beginning the trial
* Accepted method of birth control

Exclusion Criteria:

* Comorbid bipolar disorder, psychotic disorder, substance use disorder, developmental disorder or intellectual disability (IQ<70)
* Recent change (less than 4 weeks) in other medications that have potential effects on tic severity (such as alpha-2 agonists (guanfacine, clonidine or prazosin), SSRIs, clomipramine, naltrexone, lithium, anxiolytics, topiramate, baclofen etc.). Medication change is defined to include dose changes or medication discontinuation.
* Recent change in behavioral treatment for Tourette syndrome or comorbid conditions (i.e. OCD) within the last 4 weeks or initiation of behavioral therapy for tics within the last 12 weeks.
* Taking any co-medications (over the counter or prescription), food supplements/additives which can have a drug interaction with dronabinol or PEA.
* Positive pregnancy test or drug screening test
* History of cannabis dependence
* Significant Medical Comorbidity
* History of hypersensitivity to any cannabinoid or sesame oil

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dronabinol and Palmitoylethanolamide: All participants will be titrated up on Dronabinol dose during the first week of the trial (2.5mg Dronabinol for 3 days and then 5mg Dronabinol for 4 days increasing to 10mg Dronabinol for the remainder of the trial). Dronabinol will only be increased to 10mg at the week 1 assessment if the subject is tolerating the 5mg dose of Dronabinol and the Dronabinol may be reduced based on patient side-effects. All participants received two 400mg tablets of PEA daily for the same 12 weeks that they received the Dronabinol.
Period: Overall Study
Arm/Group | Dronabinol and Palmitoylethanolamide
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Dronabinol and Palmitoylethanolamide: All participants will be titrated up on Dronabinol dose during the first week of the trial (2.5mg Dronabinol for 3 days and then 5mg Dronabinol for 4 days increasing to 10mg Dronabinol for the remainder of the trial). Dronabinol will only be increased to 10mg at the week 1 assessment if the subject is tolerating the 5mg dose of Dronabinol and the Dronabinol may be reduced based on patient side-effects. Participants will be receiving PEA concomitantly.
  All participants will receive two 400mg tablets of PEA daily for the same 12 weeks that they receive the Dronabinol.
  Dronabinol: Participants will receive Dronabinol which will be slowly titrated in the first week of the study. They will be followed for a total of 12 weeks.
  Palmotoyletahnolamide: Participants will receive the PEA in a standing dose of 400mg. They will be followed for a total of 12 weeks.
Arm/Group | Dronabinol and Palmitoylethanolamide
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 35 [18 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Yale Global Severity Scale (YGTSS)Tic total score at baseline [Mean (Full Range); unit: units on a scale] — Yale Global Tic Severity Scale (YGTSS) (Total Tic Score) The YGTSS tool gives ratings in 5 domains: Total Motor Tic Score, Total Verbal Tic Score, Total Tic Score (Motor + Verbal), Overall Impairment Rating, and Global Severity Score. When calculating the Global Severity score, it is found by adding together the total motor, verbal and impairment scores. The Total Tic Severity Score has a range of 0-50, and the Global Severity Score has a range of 0- 100. A higher score on all scales suggests a more severe Tic, or a greater impact the Tic has on the person's life
  units on a scale | 38.1 [20 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Tic Severity
Description: Yale Global Tic Severity Scale (YGTSS) (Total Tic Score) The YGTSS tool gives ratings in 5 domains: Total Motor Tic Score, Total Verbal Tic Score, Total Tic Score (Motor + Verbal), Overall Impairment Rating, and Global Severity Score. When calculating the Global Severity score, it is found by adding together the total motor, verbal and impairment scores. The Total Tic Severity Score has a range of 0-50, and the Global Severity Score has a range of 0- 100. A higher score on all scales suggests a more severe Tic, or a greater impact the Tic has on the person's life.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Dronabinol and Palmitoylethanolamide: All participants will be titrated up on Dronabinol dose during the first week of the trial (2.5mg Dronabinol for 3 days and then 5mg Dronabinol for 4 days increasing to 10mg Dronabinol for the remainder of the trial). Dronabinol will only be increased to 10mg at the week 1 assessment if the subject is tolerating the 5mg dose of Dronabinol and the Dronabinol may be reduced based on patient side-effects. All participants will receive two 400mg tablets of PEA daily for the same 12 weeks that they receive the Dronabinol.
  Dronabinol: Participants will receive Dronabinol which will be slowly titrated in the first week of the study. They will be followed for a total of 12 weeks.
  Palmotoyletahnolamide: Participants will receive the PEA in a standing dose of 400mg. They will be followed for a total of 12 weeks.
Arm/Group | Dronabinol and Palmitoylethanolamide
Number analyzed (Participants) | 16
score on a scale | 7.6 [2.5 to 12.8]

ADVERSE EVENTS:
Time Frame: Collected at each study visit. Participants would come in every two weeks for twelve weeks.
Arm/Group | Dronabinol and Palmitoylethanolamide
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol and Palmitoylethanolamide (N=16)
Fatigue/Drowsiness (Nervous system disorders) | 16 (16)
Feeling "high" (Nervous system disorders) | 16 (16)
Dry Mouth (Skin and subcutaneous tissue disorders) | 15 (15)
Dizziness/Lightneadedness (Nervous system disorders) | 13 (13)
Difficulty concentrating (Nervous system disorders) | 13 (13)
Headache (Nervous system disorders) | 11 (11)
Anxiety (Psychiatric disorders) | 11 (11)
Weakness, unsteadiness (Nervous system disorders) | 11 (11)
Warmth or tingly feeling (Nervous system disorders) | 10 (10)
Gaps in memory (Nervous system disorders) | 10 (10)
Ataxia (Nervous system disorders) | 10 (10)
Clumsiness (Nervous system disorders) | 9 (9)
Lack of coordination (Nervous system disorders) | 9 (9)
Depersonalization (Nervous system disorders) | 9 (9)
Increased apetite (Metabolism and nutrition disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 8 (8)
Exagerated sense or well being (Psychiatric disorders) | 7 (7)
Red eyes (Eye disorders) | 7 (7)
Heavy limbs/muscles (Nervous system disorders) | 7 (7)
Sleep problems (insomnia) (Psychiatric disorders) | 6 (6)
Blurry vision (Eye disorders) | 6 (6)
Decrease in apetite (Metabolism and nutrition disorders) | 6 (6)
Paranoia (Psychiatric disorders) | 6 (6)
Mood changes (Psychiatric disorders) | 5 (5)
Muscle aches/pains (Musculoskeletal and connective tissue disorders) | 5 (5)
Stomach pain (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Panic attack (Psychiatric disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT03066193/Prot_SAP_000.pdf